CLINICAL TRIAL: NCT02148861
Title: A Multiple Dose Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered NNC0148-0287 (Insulin 287) in Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered NNC0148-0287 (Insulin 287) in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1436-4057; 2013-001180-22 (EudraCT Number); U1111-1140-5344 (Other: WHO)
Record Dates: First submitted 2014-04-22; First posted 2014-05-28 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin icodec; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin 287 + placebo (Experimental): Subjects will receive one of two treatment combinations: either insulin 287 + placebo or insulin degludec + placebo. Dose escalation design (4 dose levels).
  Interventions: Drug: Insulin icodec; Drug: placebo
- Insulin degludec + placebo (Active Comparator): Subjects will receive one of two treatment combinations: either insulin 287 + placebo or insulin degludec + placebo. Dose escalation design (4 dose levels).
  Interventions: Drug: insulin degludec; Drug: placebo

INTERVENTIONS:
Drug: Insulin icodec — Administered once-weekly subcutaneously (s.c., under the skin) for 35 days
  Other Names: insulin 287
  Arms: Insulin 287 + placebo
Drug: insulin degludec — Administered once-daily subcutaneously (s.c., under the skin) for 35 days
  Arms: Insulin degludec + placebo
Drug: placebo — Administered subcutaneously (s.c., under the skin) once-daily for 35 days

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of subcutaneously administered NNC0148-0287 (insulin 287) in subjects with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 18 and 64 years (both inclusive) at the time of signing informed consent
* Females of no childbearing potential [if surgically sterilized (i.e. tubal ligation, bilateral oophorectomises or hysterectomised) for at least 3 months or if post-menopausal (i.e. as defined by amenorrhoea for at least 12 months prior to screening and documented by FSH (follicle-stimulating hormone) levels above 40 U/L]
* Body mass index (BMI) between 20.0 and 35.0 kg/m^2 (both inclusive)
* Type 2 diabetes mellitus (as diagnosed clinically) for at least 12 months

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Receipt of any investigational medicinal products within 3 months before screening
* Use of oral antidiabetic drugs (OADs) or glucagon-like peptide-1 (GLP-1) receptor agonists (exenatide, liraglutide) within 3 months prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | From the first trial product administration at Day 1 until completion of the post-treatment follow-up visit (3-14 days after Visit 9, Day 65)

SECONDARY OUTCOMES:
Area under the steady-state serum insulin 287 concentration-time curve | During one dosing interval at steady-state from 0 to 168 h after last dose (Day 29)
area under the glucose infusion rate - time curve at steady-state | At Day 31 and day 35

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com